CLINICAL TRIAL: NCT00913029
Title: A Prospective, Unmasked, Randomized Evaluation of the iStent Versus Two Ocular Hypotensive Agents in Patients With Primary Open-Angle Glaucoma
Brief Title: Evaluation of the iStent Versus Two Ocular Hypotensive Agents in Patients With Primary Open-angle Glaucoma (POAG)
Acronym: SL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Second Line; Second Line Trial (Other: Glaukos)
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Eye Diseases; Glaucoma, Open-Angle; Glaucoma
Keywords: primary open angle glaucoma (POAG); OAG; glaucoma
MeSH Terms: conditions — Eye Diseases; Glaucoma, Open-Angle; Glaucoma | interventions — Stents; Latanoprost; Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stent (Active Comparator): One hundred patients will be randomized to implantation of two G2 stents in at least one eye.
  Interventions: Device: iStent
- Medication (Active Comparator): One hundred patients will be randomized to receive a fixed combination ocular hypotensive medication.
  Interventions: Drug: latanoprost/timolol

INTERVENTIONS:
Device: iStent — iStent
  Other Names: stent, Trabecular micro bypass
  Arms: Stent
Drug: latanoprost/timolol — Combination latanoprost/timolol
  Arms: Medication

SUMMARY:
Prospective, unmasked, randomized evaluation of the iStent in patients with primary open-angle glaucoma. Patients will be randomized to one of two groups: 1) iStent, or 2) medication.

DETAILED DESCRIPTION:
Two hundred patients will be enrolled in the study at up to 21 clinical sites; follow-up is through 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open-angle glaucoma
* Male or female at least 18 years of age and able to provide written informed consent
* Mean IOP (at baseline visit after washout of any medications) must be 22 mm Hg and no greater than 38 mm Hg
* Likely to be available and willing to attend follow-up visits

Exclusion Criteria:

* Angle closure glaucoma
* Secondary glaucomas
* Prior glaucoma procedures
* Elevated episcleral venous pressure from history of active thyroid orbitopathy, carotid-cavernous fistula, orbital tumors, or orbital congestive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Mean intraocular pressure (IOP) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Wells, PharmD, MBA, Study Director — Glaukos Corporation
Locations (16):
- SV Malayan Ophthalmological Center, Yerevan, Armenia
- Allgemeines Krankenhaus Wien, Vienna, Austria
- France (2):
  - CHU de Lyon Hopital Edouard Herriot, Lyon
  - CHNO des Quinze-Vingts, Paris
- Germany (3):
  - Knapschaftskrankenhaus Bochum Langendreer, Bochum
  - Helios Cliniic, Erfurt
  - Universitatsklinkum Erlangen, Erlangen
- AHEPA Hospital, Thessaloniki, Greece
- Italy (3):
  - Universita'degli Studi di Parma, Parma
  - Universita' di Torino/Dipartimento di Fisiopatologia Clinica-Clinica Oculistica, Torino
  - Azienda Ospedaliera S. Maria della Misericordia, Udine
- Military Health Service Institute, Warsaw, Poland
- Spain (3):
  - Hospital Torrevieja Salud, UTE, Alicante
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- Hinchingbrooke Hospital Moorfields, Bedford, United Kingdom

REFERENCES:
- [Result] Fea AM, Belda JI, Rekas M, Junemann A, Chang L, Pablo L, Voskanyan L, Katz LJ. Prospective unmasked randomized evaluation of the iStent inject ((R)) versus two ocular hypotensive agents in patients with primary open-angle glaucoma. Clin Ophthalmol. 2014 May 7;8:875-82. doi: 10.2147/OPTH.S59932. eCollection 2014. PMID 24855336